CLINICAL TRIAL: NCT01239693
Title: A Research Plan for a Randomised, Single-blind, Parallel Group Controlled Trial in Rural Malawi, Testing the Health Effects of Supplementing Maternal Diet During Pregnancy and Lactation and Infant Diet From 6 to 18 Months of Age With High-energy, Micronutrient Fortified Lipid-based Nutrient Supplements (LNS)
Brief Title: Supplementing Maternal and Infant Diet With High-energy, Micronutrient Fortified Lipid-based Nutrient Supplements (LNS)
Acronym: iLiNS-DYAD-M
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Kamuzu University of Health Sciences (Other); University of California, Davis (Other); Bill and Melinda Gates Foundation (Other); Finnish Institute for Health and Welfare (Other Government); University of Oulu (Other)
Responsible Party: Principal Investigator, Per Ashorn, Professor of Paediatrics, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: iLiNS-DYAD-M
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Infant Malnutrition; Malnutrition in Pregnancy
Keywords: Stunting; Growth failure; Malnutrition; Lipid based nutrient supplement; LNS; Prevention; Malawi; Sub-Saharan Africa; Dietary supplementation; Efficacy; Pregnancy; Infancy; Newborn; Child neurocognitive development; Cardiometabolic health; Lung function
MeSH Terms: conditions — Infant Nutrition Disorders; Growth Disorders; Failure to Thrive; Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IFA group (Active Comparator): Women during pregnancy: 1 tablet of iron+ folate daily until delivery (60 mg iron + 400 ug folic acid) Women during lactation (from delivery to 6 months post-partum): 1 daily tablet of calcium (200 mg), akin to placebo Children from 6 to 18 months of age: None
  Interventions: Dietary Supplement: IFA
- MMN group (Active Comparator): Women during pregnancy: 1 tablet of multiple micronutrients daily until delivery Women during lactation (from delivery to 6 months post-partum): 1 daily tablet of multiple micronutrients' Children from 6 to 18 months of age: None
  Interventions: Dietary Supplement: MMN
- LNS group (Experimental): Women during pregnancy: 1 sachet of LNS-P&L (20 g of LNS) daily until delivery Women during lactation (from delivery to 6 months post-partum): 1 daily sachet of LNS-P&L (20 g of LNS) Children from 6 to 18 months of age: 2 daily sachet of LNS-20gM (20 g of LNS)
  Interventions: Dietary Supplement: LNS

INTERVENTIONS:
Dietary Supplement: IFA — Women during pregnancy: 1 tablet of iron+ folate daily until delivery (60 mg iron + 400 ug folic acid) Women during lactation (from delivery to 6 months post-partum): 1 daily tablet of calcium (200 mg), akin to placebo Children from 6 to 18 months of age: None
  Arms: IFA group
Dietary Supplement: MMN — Women during pregnancy: 1 tablet of multiple micronutrients daily until delivery Women during lactation (from delivery to 6 months post-partum): 1 daily tablet of multiple micronutrients Children from 6 to 18 months of age: None
  Arms: MMN group
Dietary Supplement: LNS — Women during pregnancy: 1 sachet of LNS-P&L (20 g of LNS) daily until delivery Women during lactation (from delivery to 6 months post-partum): 1 daily sachet of LNS-P&L (20 g of LNS) Children from 6 to 18 months of age: 2 daily sachet of LNS-20gM (20 g of LNS)
  Arms: LNS group

SUMMARY:
The use of lipid-based nutrients (LNS), such as Nutributter or fortified spread (FS), have been associated with improved growth and development outcomes among infants in Ghana and Malawi. Modified versions of such supplements have been developed to improve their nutrient density and quality and to lower their costs. Such modified products have proven acceptable to pregnant women in Malawi and Ghana. In the present trial, the investigators aim to test the effect of LNS on pregnancy and child outcomes, when given during pregnant and lactating women and their infants from 6 to 18 months of age. In control groups, participants will receive either iron+folate tables during pregnancy only or multiple micronutrient tablets during pregnancy and first six months of lactations. The main hypothesis to be tested suggests that the mean length-for-age Z-score (LAZ) of 18-month-old infants who received LNS between 6 and 18 months of age and whose mothers were provided with LNS during pregnancy and the first 6 months of lactation is higher than the mean LAZ score of same age infants who received no dietary supplements and whose mothers received iron-folate supplementation during pregnancy only.

To detect the long-term effect of the LNS supplementation, we now propose to conduct a follow-up study when the children are 9 years old, to see if the intervention had effect on children's growth, cardiometabolic and respiratory status and neurocognitive development.

DETAILED DESCRIPTION:
Pregnant women will be identified from the antenatal clinics of 4 governmental and 2 other health centres. A total of 1400 women meeting set criteria will be randomised into receiving one of the following interventions: 1) Iron and folic acid supplementation to the mother during pregnancy only (IFA group), 2). Multiple micronutrient supplementation to the mother during pregnancy and six months thereafter (MMN group), 3) Lipid-based nutrient supplements to the mother during pregnancy and six months thereafter and to the child from 6 to 18 months of age (LNS group).

The mothers will receive LNS or the multiple micronutrients at 2-weekly intervals at their homes during pregnancy and weekly during first six months of lactation. Children in the LNS group will receive LNS weekly, starting at 6 months. Mothers will be medically examined and tested for defined laboratory parameters at enrolment, at 36 gestation weeks, at birth or soon thereafter, and at 6 months after delivery. Child size will be assessed at birth or soon thereafter and at 3, 6, 12, and 18 months of age. The mothers will undergo a morbidity evaluation fortnightly and the children weekly.

864 mother-infant pairs will undergo the complete intervention and follow-up, as described above. The remaining 536 participants will undergo a simplified intervention and follow-up, in which there are no interventions after birth and the child follow-up consists only of 4 3 health centre and one home visits; first at 1 week, then at six weeks (at home) and at 6 and 18 months of age.

A sub-study on the the development of intestinal microbiome was added in August 2011. This entails the collection of stool samples from the mother at 1 month after delivery, breast milk samples from the mothers at 1, 3, and 6 months after delivery and stool and urine samples from the children repeated during the a8 months of intervention. The aim of this subproject is to study the development of the infants' intestinal microbiota, its predictors and its association to child growth and other health outcomes. At the same time point, the sample size was reduced from 2400 to 1400 participants (due to constraints in funding).

A one year post-intervention follow-up for participants in the complete follow-up was added to the study protocol in August 2013. The intervention will be stopped when the participants are 18 months old. Thereafter, there will be an anthropometrirc assessment and blood and urine draw at the study clinic at 24 and 30 months of age. Stool samples will be collected from the participants at the age of 21, 24, 27 and 30 months, to study the development of intestinal microbiome.

In a follow-up study, when the children are 10 years old, we will assess:

1. child growth using standard anthropometric measures,
2. cardiometabolic health by measuring body composition, blood pressure and plasma lipids,
3. neurodevelopment by measuring neural function, cognitive skills and education attainment using EE and EGMA and Raven's questionnaires,
4. lung function with spirometry and allergy symptoms and asthma using ISAAC questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound confirmed pregnancy of no more than 20 completed gestation weeks
* Permanent resident of Mangochi District Hospital, Malindi Hospital or Lungwena Health Centre catchment areas
* Availability during the period of the study
* Signed informed consent

Exclusion Criteria:

* Less than 15 years of age
* Need for frequent medical attention due to a chronic health condition
* Diagnosed asthma treated with regular medication
* Severe illness warranting hospital referral
* History of allergy towards peanuts
* History of anaphylaxis or serious allergic reaction to any substance, requiring emergency medical care
* Pregnancy complications evident at enrolment visit (moderate to severe oedema, blood Hb concentration < 5 g / dl, systolic blood pressure (BP) > 160 mmHg or diastolic BP > 100 mmHg)
* Earlier participation in the iLiNS-DYAD-M trial
* Concurrent participation in any other clinical trial

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1391 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Birth weight | approx 20 weeks after enrollment (within 48 hours)
Newborn length | At 1 week of age
Length for age Z-score (LAZ) at 18 months of age | 12 months after enrollment (age 18 months)

SECONDARY OUTCOMES:
Anthropometric status (weight, BMI, mid upper arm circumference and triceps and sub-scapular skin-fold thickness) | at ~ 36 wk gestation and 6 months postpartum
Gestational age at delivery, proportion of preterm deliveries | At delivery
Proportion of low birth weight babies | At birth
Anaemia and iron status (Hb, ZPP, transferrin receptor), other micronutrient status (vitamin A, B-vitamins, zinc), malarial antigen | At ~ 36 wk gestation and 6 mo postpartum
Red blood cell essential fatty acid status | At ~ 36 wk gestation
Urinary iodine | At ~ 36 wk gestation
Total plasma cholesterol concentration | At ~ 36 wk gestation
Basal salivary cortisol concentration | At ~ 28 and ~ 36 wk gestation
Blood pressure | At 36 wk gestation
Breast milk composition (essential fatty acids, vitamin A, B-vitamins) | At 6 mo postpartum
Depressive symptoms (which may be related to essential fatty acid status) | At 4 weeks and at 6 months postpartum
Incidence of febrile malaria episodes | During pregnancy
Peripheral blood malaria parasitaemia | At 32 wk gestation and at delivery
Placental malaria histology | At delivery
Evidence of defined bacteria in the chorionic membranes at delivery (quantitative DNA amplification method) | At birth
Prevalence of Neisseria gonorrhoea, Chlamydia trachomatis, in swab samples taken from maternal uterine cervix(qualitative DNA amplification method) | At one week after delivery
Prevalence of bacterial vaginosis, Trichomonas vaginalis, or candidiasis, in swab samples taken from maternal vagina(direct microscopy) | At one week after delivery
Malaria immunity | At enrolment, at ~ 36 wk gestation, and 6 months post-partum
Anthropometric infant status (weight, length, head circumference and mid upper arm circumference) | At 7 days of age and at 6, 12 and 18 months of age. After the intervention at 24 and 30 months and at 10 y of age.
Infant anaemia and iron status (Hb, ZPP), micronutrient (vitamin A, B-vitamins) and essential fatty acids status, evidence of acute inflammation (CRP, AGP), and malarial antigen and microscopy | At 6 and 18 months of age
Incidence of neonatal hospitalizations | At or before age 28 days
Clinical morbidity | Between 0 and 18 months of age
Child feeding practices and maternal report of child sleep patterns | At 6, 12 and 18 months of age
Antibody response to measles vaccination | At 18 months of age
Malaria immunity | At 6 and 18 months of age
Basal salivary cortisol concentration | At 6, 12 and 18 months of age
Cortisol response to acute stress | At 6 and 18 months of age
Achievement of five motor milestones and four other developmental milestones | From 0 to 18 mo
Neurobehavioral development | At 18 months of age
Incidence of serious adverse events | During pregnancy and 18 months of infant follow-up
Prevalence of maternal periodontitis | At one week after delivery
Maternal cognition | 6 months after delivery
  Measured with several different tests
Mother - child interaction | 6 months after delivery
  Measured with a number of observational tests and questionnaires
The composition of intestinal microbiota | 1, 2, 3, 4, 5, 6, 9, 12, 15, 18, 21, 24, 27, and 30 months of child age
  Done with 16s sequencing, from stored stool samples
diastolic blood pressure | Child is 10 years
  Mobil-o-Graph blood pressure monitoring system
central blood pressure | Child is 10 years
  Mobil-o-Graph blood pressure monitoring system
pulse rate | Child is 10 years
  Mobil-o-Graph blood pressure monitoring system
vascular resistance | Child is 10 years
  Mobil-o-Graph blood pressure monitoring system
plasma concentration of glucose | Child is 10 years
  Cobas c702 machine
plasma concentration of cholesterol | Child is 10 years
  Cobas c702 machine
plasma concentration of HDL/LDL cholesterol | Child is 10 years
  Cobas c702 machine
plasma concentration of triglycerides | Child is 10 years
  Cobas c702 machine
plasma concentration of c-reactive protein | Child is 10 years
  Cobas c702 machine
plasma concentration of alkaline phosphatase | Child is 10 years
  Cobas c702 machine
plasma concentration of aspartyl alanine transferase | Child is 10 years
  Cobas c702 machine
plasma concentration of potassium | Child is 10 years
  Cobas c702 machine
plasma concentration of sodium | Child is 10 years
  Cobas c702 machine
plasma concentration of urate | Child is 10 years
  Cobas c702 machine
Spirometry measures functional volume of the lungs | Child is 10 years
  Global Lung Function Initiative standards, Medikro pro spirometry
asthma symptoms | Child is 10 years
  ISAAC questionnaire
allergy symptoms | Child is 10 years
  ISAAC questionnaire
neural functioning | Child is 10 years
  EEG
processing speed | Child is 10 years
  EEG
oculomotor reaction time | Child is 10 years
  eye-tracking
academic achievement | Child is 10 years
  Early Grade Mathematics Assessment, EGMA
height | Child is 10 years
sitting height | Child is 10 years
weight | Child is 10 years
head circumference | Child is 10 years
mid-upper arm circumference | Child is 10 years
body composition | Child is 10 years
  Tanita MC-780 MAS

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Principal Investigator — University of Tampere Medical School
Locations (1):
- University of Malawi, College of Medicine, Mangochi, Malawi

REFERENCES:
- [Derived] Adu-Afarwuah S, Arnold CD, Lartey A, Okronipa H, Maleta K, Ashorn P, Ashorn U, Dewey KG. Prevalence of morbidity symptoms among pregnant and postpartum women receiving different nutrient supplements in Ghana and Malawi: A secondary outcome analysis of two randomised controlled trials. Matern Child Nutr. 2023 Jul;19(3):e13501. doi: 10.1111/mcn.13501. Epub 2023 Apr 6. PMID 37021807
- [Derived] Liu Z, Fan YM, Ashorn P, Chingwanda C, Maleta K, Hallamaa L, Hyoty H, Chaima D, Ashorn U. Lack of Associations between Environmental Exposures and Environmental Enteric Dysfunction among 18-Month-Old Children in Rural Malawi. Int J Environ Res Public Health. 2022 Sep 1;19(17):10891. doi: 10.3390/ijerph191710891. PMID 36078607
- [Derived] Salenius M, Pyykko J, Ashorn U, Dewey KG, Gondwe A, Harjunmaa U, Maleta K, Nkhoma M, Vosti SA, Ashorn P, Adubra L. Association between prenatal provision of lipid-based nutrient supplements and caesarean delivery: Findings from a randomised controlled trial in Malawi. Matern Child Nutr. 2022 Oct;18(4):e13414. doi: 10.1111/mcn.13414. Epub 2022 Jul 31. PMID 35909334
- [Derived] Haskell MJ, Maleta K, Arnold CD, Jorgensen JM, Fan YM, Ashorn U, Matchado A, Monangi NK, Zhang G, Xu H, Belling E, Landero J, Chappell J, Muglia LJ, Hallman M, Ashorn P, Dewey KG. Provision of Small-Quantity Lipid-Based Nutrient Supplements Increases Plasma Selenium Concentration in Pregnant Women in Malawi: A Secondary Outcome of a Randomized Controlled Trial. Curr Dev Nutr. 2022 Mar 7;6(3):nzac013. doi: 10.1093/cdn/nzac013. eCollection 2022 Mar. PMID 35317414
- [Derived] Smith JW, Matchado AJ, Wu LS, Arnold CD, Burke SM, Maleta KM, Ashorn P, Stewart CP, Shaikh S, Ali H, Labrique AB, West KP Jr, Christian P, Dewey KG, Groopman JD, Schulze KJ. Longitudinal Assessment of Prenatal, Perinatal, and Early-Life Aflatoxin B1 Exposure in 828 Mother-Child Dyads from Bangladesh and Malawi. Curr Dev Nutr. 2022 Jan 7;6(2):nzab153. doi: 10.1093/cdn/nzab153. eCollection 2022 Feb. PMID 35155983
- [Derived] Kortekangas E, Fan YM, Chaima D, Lehto KM, Malamba-Banda C, Matchado A, Chingwanda C, Liu Z, Ashorn U, Cheung YB, Dewey KG, Maleta K, Ashorn P. Associations between Gut Microbiota and Intestinal Inflammation, Permeability and Damage in Young Malawian Children. J Trop Pediatr. 2022 Feb 3;68(2):fmac012. doi: 10.1093/tropej/fmac012. PMID 35149871
- [Derived] Adu-Afarwuah S, Arnold CD, Lartey A, Okronipa H, Maleta K, Ashorn P, Ashorn U, Fan YM, Matchado A, Kortekangas E, Oaks BM, Jackson KH, Dewey KG. Small-Quantity Lipid-Based Nutrient Supplements Increase Infants' Plasma Essential Fatty Acid Levels in Ghana and Malawi: A Secondary Outcome Analysis of the iLiNS-DYAD Randomized Trials. J Nutr. 2022 Jan 11;152(1):286-301. doi: 10.1093/jn/nxab329. PMID 34543432
- [Derived] Jorgensen JM, Young R, Ashorn P, Ashorn U, Chaima D, Davis JCC, Goonatilleke E, Kumwenda C, Lebrilla CB, Maleta K, Sadalaki J, Totten SM, Wu LD, Zivkovic AM, Dewey KG. Associations of Human Milk Oligosaccharides and Bioactive Proteins with Infant Morbidity and Inflammation in Malawian Mother-Infant Dyads. Curr Dev Nutr. 2021 Apr 29;5(5):nzab072. doi: 10.1093/cdn/nzab072. eCollection 2021 May. PMID 34084993
- [Derived] Jorgensen JM, Young R, Ashorn P, Ashorn U, Chaima D, Davis JCC, Goonatilleke E, Kumwenda C, Lebrilla CB, Maleta K, Prado EL, Sadalaki J, Totten SM, Wu LD, Zivkovic AM, Dewey KG. Associations of human milk oligosaccharides and bioactive proteins with infant growth and development among Malawian mother-infant dyads. Am J Clin Nutr. 2021 Jan 4;113(1):209-220. doi: 10.1093/ajcn/nqaa272. PMID 33096556
- [Derived] Adu-Afarwuah S, Arnold CD, Maleta K, Ashorn P, Ashorn U, Jorgensen JM, Fan YM, Nkhoma M, Bendabenda J, Matchado A, Dewey KG. Consumption of multiple micronutrients or small-quantity lipid-based nutrient supplements containing iodine at the recommended dose during pregnancy, compared with iron and folic acid, does not affect women's urinary iodine concentration in rural Malawi: a secondary outcome analysis of the iLiNS DYAD trial. Public Health Nutr. 2021 Jul;24(10):3049-3057. doi: 10.1017/S1368980020003250. Epub 2020 Oct 15. PMID 33054890
- [Derived] Kamng'ona AW, Young R, Arnold CD, Patson N, Jorgensen JM, Kortekangas E, Chaima D, Malamba C, Ashorn U, Cheung YB, Ashorn P, Maleta K, Dewey KG. Provision of Lipid-Based Nutrient Supplements to Mothers During Pregnancy and 6 Months Postpartum and to Their Infants from 6 to 18 Months Promotes Infant Gut Microbiota Diversity at 18 Months of Age but Not Microbiota Maturation in a Rural Malawian Setting: Secondary Outcomes of a Randomized Trial. J Nutr. 2020 Apr 1;150(4):918-928. doi: 10.1093/jn/nxz298. PMID 31909811
- [Derived] Kortekangas E, Young R, Cheung YB, Fan YM, Jorgensen JM, Kamng'ona AW, Chaima D, Ashorn U, Dewey KG, Maleta K, Ashorn P. A Prospective Study on Child Morbidity and Gut Microbiota in Rural Malawi. J Pediatr Gastroenterol Nutr. 2019 Oct;69(4):431-437. doi: 10.1097/MPG.0000000000002435. PMID 31436705
- [Derived] Bendabenda J, Patson N, Hallamaa L, Ashorn U, Dewey KG, Ashorn P, Maleta K. Does anthropometric status at 6 months predict the over-dispersion of malaria infections in children aged 6-18 months? A prospective cohort study. Malar J. 2019 Apr 22;18(1):143. doi: 10.1186/s12936-019-2778-y. PMID 31010435
- [Derived] Barua P, Beeson JG, Maleta K, Ashorn P, Rogerson SJ. The impact of early life exposure to Plasmodium falciparum on the development of naturally acquired immunity to malaria in young Malawian children. Malar J. 2019 Jan 18;18(1):11. doi: 10.1186/s12936-019-2647-8. PMID 30658632
- [Derived] Oaks BM, Jorgensen JM, Baldiviez LM, Adu-Afarwuah S, Maleta K, Okronipa H, Sadalaki J, Lartey A, Ashorn P, Ashorn U, Vosti S, Allen LH, Dewey KG. Prenatal Iron Deficiency and Replete Iron Status Are Associated with Adverse Birth Outcomes, but Associations Differ in Ghana and Malawi. J Nutr. 2019 Mar 1;149(3):513-521. doi: 10.1093/jn/nxy278. PMID 30629202
- [Derived] Bendabenda J, Patson N, Hallamaa L, Mbotwa J, Mangani C, Phuka J, Prado EL, Cheung YB, Ashorn U, Dewey KG, Ashorn P, Maleta K. The association of malaria morbidity with linear growth, hemoglobin, iron status, and development in young Malawian children: a prospective cohort study. BMC Pediatr. 2018 Dec 28;18(1):396. doi: 10.1186/s12887-018-1378-2. PMID 30593271
- [Derived] Barua P, Chandrasiri UP, Beeson JG, Dewey KG, Maleta K, Ashorn P, Rogerson SJ. Effect of nutrient supplementation on the acquisition of humoral immunity to Plasmodium falciparum in young Malawian children. Malar J. 2018 Feb 7;17(1):74. doi: 10.1186/s12936-018-2224-6. PMID 29415730
- [Derived] Doyle R, Gondwe A, Fan YM, Maleta K, Ashorn P, Klein N, Harris K. A Lactobacillus-Deficient Vaginal Microbiota Dominates Postpartum Women in Rural Malawi. Appl Environ Microbiol. 2018 Mar 1;84(6):e02150-17. doi: 10.1128/AEM.02150-17. Print 2018 Mar 15. PMID 29305501
- [Derived] Adams KP, Ayifah E, Phiri TE, Mridha MK, Adu-Afarwuah S, Arimond M, Arnold CD, Cummins J, Hussain S, Kumwenda C, Matias SL, Ashorn U, Lartey A, Maleta KM, Vosti SA, Dewey KG. Maternal and Child Supplementation with Lipid-Based Nutrient Supplements, but Not Child Supplementation Alone, Decreases Self-Reported Household Food Insecurity in Some Settings. J Nutr. 2017 Dec;147(12):2309-2318. doi: 10.3945/jn.117.257386. Epub 2017 Oct 4. PMID 28978680
- [Derived] Jorgensen JM, Arnold C, Ashorn P, Ashorn U, Chaima D, Cheung YB, Davis JC, Fan YM, Goonatilleke E, Kortekangas E, Kumwenda C, Lebrilla CB, Maleta K, Totten SM, Wu LD, Dewey KG. Lipid-Based Nutrient Supplements During Pregnancy and Lactation Did Not Affect Human Milk Oligosaccharides and Bioactive Proteins in a Randomized Trial. J Nutr. 2017 Oct 1;147(10):1867-1874. doi: 10.3945/jn.117.252981. PMID 28794206
- [Derived] Oaks BM, Young RR, Adu-Afarwuah S, Ashorn U, Jackson KH, Lartey A, Maleta K, Okronipa H, Sadalaki J, Baldiviez LM, Shahab-Ferdows S, Ashorn P, Dewey KG. Effects of a lipid-based nutrient supplement during pregnancy and lactation on maternal plasma fatty acid status and lipid profile: Results of two randomized controlled trials. Prostaglandins Leukot Essent Fatty Acids. 2017 Feb;117:28-35. doi: 10.1016/j.plefa.2017.01.007. Epub 2017 Jan 25. PMID 28237085
- [Derived] Nkhoma M, Ashorn P, Ashorn U, Dewey KG, Gondwe A, Mbotwa J, Rogerson S, Taylor SM, Maleta K. Providing lipid-based nutrient supplement during pregnancy does not reduce the risk of maternal P falciparum parasitaemia and reproductive tract infections: a randomised controlled trial. BMC Pregnancy Childbirth. 2017 Jan 17;17(1):35. doi: 10.1186/s12884-016-1215-2. PMID 28095801
- [Derived] Chandrasiri UP, Fowkes FJ, Beeson JG, Richards JS, Kamiza S, Maleta K, Ashorn P, Rogerson SJ. Association between malaria immunity and pregnancy outcomes among Malawian pregnant women receiving nutrient supplementation. Malar J. 2016 Nov 9;15(1):547. doi: 10.1186/s12936-016-1597-7. PMID 27829430
- [Derived] Klevor MK, Adu-Afarwuah S, Ashorn P, Arimond M, Dewey KG, Lartey A, Maleta K, Phiri N, Pyykko J, Zeilani M, Ashorn U. A mixed method study exploring adherence to and acceptability of small quantity lipid-based nutrient supplements (SQ-LNS) among pregnant and lactating women in Ghana and Malawi. BMC Pregnancy Childbirth. 2016 Aug 30;16(1):253. doi: 10.1186/s12884-016-1039-0. PMID 27577112
- [Derived] Prado EL, Abbeddou S, Adu-Afarwuah S, Arimond M, Ashorn P, Ashorn U, Brown KH, Hess SY, Lartey A, Maleta K, Ocansey E, Ouedraogo JB, Phuka J, Some JW, Vosti SA, Yakes Jimenez E, Dewey KG. Linear Growth and Child Development in Burkina Faso, Ghana, and Malawi. Pediatrics. 2016 Aug;138(2):e20154698. doi: 10.1542/peds.2015-4698. PMID 27474016
- [Derived] Prado EL, Maleta K, Ashorn P, Ashorn U, Vosti SA, Sadalaki J, Dewey KG. Effects of maternal and child lipid-based nutrient supplements on infant development: a randomized trial in Malawi. Am J Clin Nutr. 2016 Mar;103(3):784-93. doi: 10.3945/ajcn.115.114579. Epub 2016 Feb 3. PMID 26843155
- [Derived] Stewart CP, Oaks BM, Laugero KD, Ashorn U, Harjunmaa U, Kumwenda C, Chaima D, Maleta K, Ashorn P, Dewey KG. Maternal cortisol and stress are associated with birth outcomes, but are not affected by lipid-based nutrient supplements during pregnancy: an analysis of data from a randomized controlled trial in rural Malawi. BMC Pregnancy Childbirth. 2015 Dec 22;15:346. doi: 10.1186/s12884-015-0793-8. PMID 26694646
- [Derived] Chandrasiri UP, Fowkes FJ, Richards JS, Langer C, Fan YM, Taylor SM, Beeson JG, Dewey KG, Maleta K, Ashorn P, Rogerson SJ. The impact of lipid-based nutrient supplementation on anti-malarial antibodies in pregnant women in a randomized controlled trial. Malar J. 2015 May 10;14:193. doi: 10.1186/s12936-015-0707-2. PMID 25957793
- [Derived] Ashorn P, Alho L, Ashorn U, Cheung YB, Dewey KG, Gondwe A, Harjunmaa U, Lartey A, Phiri N, Phiri TE, Vosti SA, Zeilani M, Maleta K. Supplementation of Maternal Diets during Pregnancy and for 6 Months Postpartum and Infant Diets Thereafter with Small-Quantity Lipid-Based Nutrient Supplements Does Not Promote Child Growth by 18 Months of Age in Rural Malawi: A Randomized Controlled Trial. J Nutr. 2015 Jun;145(6):1345-53. doi: 10.3945/jn.114.207225. Epub 2015 Apr 29. PMID 25926413
- [Derived] Ashorn P, Alho L, Ashorn U, Cheung YB, Dewey KG, Harjunmaa U, Lartey A, Nkhoma M, Phiri N, Phuka J, Vosti SA, Zeilani M, Maleta K. The impact of lipid-based nutrient supplement provision to pregnant women on newborn size in rural Malawi: a randomized controlled trial. Am J Clin Nutr. 2015 Feb;101(2):387-97. doi: 10.3945/ajcn.114.088617. Epub 2014 Dec 10. PMID 25646337
- See also: College of Medicine homepage — http://www.medcol.mw/
- See also: Publication on the primary birth outcome results — http://www.ncbi.nlm.nih.gov/pubmed/25646337
- See also: Publication on the primary child growth outcome results — http://www.ncbi.nlm.nih.gov/pubmed/25926413